CLINICAL TRIAL: NCT03294837
Title: Treatment of Ventilator Associated Pneumonia in Pediatric Intensive Care Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, yostina ramzy, doctor, Assiut University
Other Study IDs: treatment of VAP in picu
Record Dates: First submitted 2017-09-16; First posted 2017-09-27 (Actual); Last update posted 2017-09-27 (Actual); Status verified 2017-09

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
treatment of ventilator associated pneumonia in pediatric intensive care unit according to the American guidelines

DETAILED DESCRIPTION:
to assess the degree of adherence of pediatric physicians of assiut university children hospital to the American guidelines of treatment of ventilator associated pneumonia in pediatric intensive care unit searching for defects,obstacles,or need to improve health service.

ELIGIBILITY:
Inclusion Criteria:

- Children of both sexes. - Aged from 1 month to 18 years. - The patients are fulfilling the diagnostic criteria of ventilator associated pneumonia.

Exclusion Criteria:

- Patients aged less than 1 month. - Patients who are intubated and mechanically ventilated for less than 48 hours.

Ages: 1 Month to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: to assess the degree of adherence of pediatric physicians of assiut university children hospital to the american guidelines of treatment of ventilator associated pneumonia in pediatric intensive care unit.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
treatment of ventilator associated pneumonia in pediatric intensive care unit | 9 month - 1 year
  to assess the quality of care and treatment of ventilator associated pneumonia in pediatric intensive care unit in assiut university children hospital according to the american guidelines and evaluation of the performance of the unit as regard sticking to the guidelines of treatment of VAP

REFERENCES:
- [Background] Chang I, Schibler A. Ventilator Associated Pneumonia in Children. Paediatr Respir Rev. 2016 Sep;20:10-16. doi: 10.1016/j.prrv.2015.09.005. Epub 2015 Sep 25. PMID 26527358
- [Background] Amanati A, Karimi A, Fahimzad A, Shamshiri AR, Fallah F, Mahdavi A, Talebian M. Incidence of Ventilator-Associated Pneumonia in Critically Ill Children Undergoing Mechanical Ventilation in Pediatric Intensive Care Unit. Children (Basel). 2017 Jul 3;4(7):56. doi: 10.3390/children4070056. PMID 28671616